



#### SOWA-ICU

Signs and symptoms of opioid-associated iatrogenic withdrawal in critically ill adults

RESEARCH PROTOCOL

Pharmacy Residents:
Laura Delucilla, PharmD, MSc Candidate

Jean-François Cabot, PharmD, MSc candidate

Qian Li, PharmD, MSc candidate

Karima Zerrouki, PharmD, MSc candidate

McGill University Health Centre

Research Director/Investigator:

Marc Perreault, PharmD, MSc, FCSHP

Clinical Directors:

Marie-Soleil Delisle, PharmD, MSc

Marc Alexandre Duceppe, PharmD, MSc

Collaborators

Leon Tourian, MD, Psychiatrist, MGH

Dev Jayaraman, MD, Intensivist, MGH

Sulaiman Khadadah, ICU Fellow

Celine Gélinas, RN, PhD, JGH

Lisa Burry, PharmD, Mount Sinai, Toronto

PHA6220 – Research in Pharmacy

Master in Advanced Pharmacotherapy

Faculty of Pharmacy

December 1st, 2017

Version 4 Date: April 4th 2018

# **Table of Contents**

| 1. | Introduction | 1 |
|---|---|---|
| 2. | Literature review | 1 |
| 3. | Research objectives | 3 |
| | Methods | 344555 |
| 5. | Data analysis 5.1 Statistical analysis 5.1.1 Descriptive statistics 5.1.2 Statistical inference 5.2 Sample size | <b>11</b><br>11 |
| 6. | Advantages and limitations | 11 |
| 7. | Relevance of study | . 12 |
| 8. | Ethical considerations and patient consent | . 12 |
| 9. | References | . 14 |
| | ). Time frame and budget | |
| 11 | Appendix I. Research strategy in Medline | 19<br>21<br>id<br>27<br>ed<br>28<br>29 |
| | Appendix X. Richmond Agitation-Sedation Scale (RASS) developed by Sessler et al | |

| Appendix XI. Agitated Behavior Scale (ABS) developed by Carrigan et al | 34 |
|---|---|
| Appendix XII. Critical-Care Pain Observation Tool (CPOT) developed by Ge | elinas et al35 |
| Appendix XIII. Numeric Rating Scale (NRS) | 36 |

# **Abbreviation list**

ICU Intensive care unit

IWS Iatrogenic withdrawal syndrome
MGH Montreal General Hospital
MUHC McGill University Health Centre

OIWS Opioid-associated introgenic withdrawal syndrome

PICU Pediatric intensive care unit RVH Royal Victoria Hospital

Version 4 Date: April 4 2018

#### 1. Introduction

Adult medical, surgical and trauma intensive care unit (ICU) patients routinely experience pain, agitation, delirium and anxiety (1). Opioids and benzodiazepines are the primary medications to relieve pain, facilitate mechanical ventilation and decrease physiological and psychological stress in the critically ill (1). In a prospective, observational study in 51 Canadian ICUs, 92% of patients received opioids and sedatives at least once during mechanical ventilation (2). Upon repeated and prolonged administration, opioid tolerance may develop as a result of receptor desensitization and upregulation of excitatory intracellular pathways (2, 3). When these drugs are abruptly discontinued or rapidly tapered, patients may develop a cluster of signs and symptoms known as the acute iatrogenic withdrawal syndrome (IWS). While this phenomenon is well described in the pediatric critical care population, there is a paucity of data in critically ill adults (4-7). IWS has been associated with negative clinical outcomes such as increased length of hospital stays, prolonged duration of mechanical ventilation and higher cost of hospitalization (4-7).

In one prospective, observational study, the reported incidence of IWS in the adult ICU population was 16.7% (8). In prospective studies done in the pediatric ICU (PICU), observed incidence was 7.5 to 100% (9). Two assessment tools have been validated in children: The Withdrawal Assessment Tool-Version 1 (WAT-1) and the Sophia Observation Withdrawal Symptoms-scale (SOS) (10). No such tool currently exists in the adult ICU (9).

Identifying IWS can be challenging in the critically ill. Several confounding factors (delirium, worsening of critical illness, presence of multiple agents with potential to cause withdrawal, comorbidities) may mimic symptoms similar to opioid or benzodiazepine withdrawal (6, 11). To our knowledge, no study on the symptomatology of IWS has been conducted to describe opioid or benzodiazepine withdrawal exclusively. This is most likely due to the presentation similarities of both syndromes and frequent concomitant use of these drugs in the ICU setting (4, 9).

No physiological markers have been identified to correlate with IWS. In outpatients with chronic opioid addiction, several studies have shown a significant association between increased cortisol and catecholamine levels and acute withdrawal following naloxone reversal. Cortisol and catecholamines are two stress markers that reflect the state of distress and adrenergic hyperstimulation characteristic of opioid withdrawal (12).

To date, the clinical presentation of opioid withdrawal in the adult ICU has not been characterized in a prospective setting. The present study thus aims to describe the symptomatology of opioid-associated iatrogenic withdrawal in two adult tertiary care centers in Montréal, Québec, Canada and explore the potential of using serum cortisol as a biomarker (4, 9).

#### 2. Literature review

Research strategy can be found in Appendix I.

### Epidemiology

A systematic review on the epidemiology, risk factors and symptomatology of IWS was recently conducted and identified only one prospective study on IWS in the adult ICU population, which reported an incidence of 16.7% (8, 9). In retrospective trials, incidence ranged from 19.7 to 100% (9). These heterogeneous results are likely attributed to the lack of standardized definition and evaluation of IWS (9).

#### Risk factors

There is significant overlap in the IWS risk factors identified in pediatric and adult populations such as younger age (3, 4, 7, 9) duration of continuous opioid therapy (i.e. more than three to five days) and prolonged benzodiazepine exposure (4, 5, 7, 9, 13-17). Additional risk factors identified specifically in the adult ICU include higher daily doses of opioids and benzodiazepines, as well as the presence of acute respiratory distress syndrome (ARDS) (7, 9). In the PICU, prolonged exposure prior to weaning


and total cumulative opioid and benzodiazepine doses have been associated with an increased risk of IWS (4, 5, 14, 15). The onset of withdrawal symptoms can occur within 12 hours following opioid discontinuation and may be precipitated by an abrupt taper or the administration of opioid antagonists (1, 18).

#### Clinical presentation

Most literature is extracted from PICU studies designed with the objective of developing or validating IWS assessment tools (16). Ista et al. compiled a list of 26 symptoms of mixed withdrawal as reported in the literature and evaluated the co-occurrence of IWS symptoms in low and high risk patients (19). An expert panel identified 15 symptoms encompassing the central nervous system (anxiety, agitation, inconsolable crying, grimacing, sleep disturbance, hallucinations), autonomic dysfunction (increased muscle tension, muscle twitching, tremors, tachycardia, tachypnea, fever, sweating) and gastrointestinal problems (vomiting, diarrhea) (19, 20). However, the investigators did not control for potential confounders of IWS diagnosis such as inadequate pain management or delirium. A review by Chiu et al. identified symptoms of opioid withdrawal specific to the neonatal and PICU populations such as inconsolable crying, irritability, grimacing, tremors, increased muscle tone, poor feeding, vomiting, diarrhea, sleep disturbance, hyperactive Moro reflex, fever, nasal stuffiness, sweating and yawning (4). However, evaluation of symptoms and outcomes were done by the same practitioner in select studies, which may have confounded the results (4, 21).

Opioid withdrawal appears to present differently in adults (4). In a prospective study evaluating the validity of the WAT-1 in the adult ICU, commonly observed symptoms in the PICU such as diarrhea, vomiting and fever did not correlate with a diagnosis of IWS (8, 22). Chiu et al. reports that withdrawal symptoms in adults tend to begin with anxiety, irritability, agitation and dysphoria, followed by sweating, rhinorrhea, tachypnea, insomnia and yawning in the acute phase. Symptoms such as mydriasis, tachycardia, hypertension, nausea, vomiting, piloerection and fever manifest during subsequent phases of withdrawal (4). In the retrospective study by Cammarano et al., IWS was diagnosed using a modified Himmelsbach scale, which assesses the severity of opioid withdrawal in chronic users only (7, 23). Thus, the symptoms identified in this study may not be applicable to opioid-naive patients. It is currently unclear whether all these symptoms can be identified in opioid-naive critically ill patients

The distinction between opioid and benzodiazepine withdrawal remains unclear because both drugs are often used simultaneously in the ICU setting. Duceppe et al. reports that there are currently no adult or pediatric ICU studies that evaluated the incidence of isolated opioid or benzodiazepine withdrawal symptoms (9). The 2002 adult critical care guidelines, updated in 2013, identifies nausea, vomiting, sweating, agitation, restlessness, irritability, anxiety and muscle cramps as common symptoms to both acute opioid and benzodiazepine withdrawal (1, 18). Benzodiazepine and opioid withdrawal symptoms largely overlap, which contributes to the difficulty in describing both syndromes adequately (20, 24).

#### Assessment tools

As stated previously, in the PICU, two validated tools are commonly used to assess IWS: the WAT-1 and the SOS. Both are included in the 2016 European clinical guidelines for pain, sedation, withdrawal and delirium assessment in critically ill infants and children (10). However, they were validated in a manner that could potentially affect the results' reliability – in the psychometric evaluation studies, the same nurse scored both the tool and withdrawal severity. The lack of blinding to the presence of IWS and the lack of independent evaluation thus-make those studies susceptible to observer bias. The WAT-1 performed poorly in the adult ICU, suggesting that the presentation of IWS is different in adults as compared to children (4).

#### **Biomarkers**

The literature on opioid dependence has consistently demonstrated elevated levels of cortisol (12, 25-38) and catecholamines (12, 39-43) during the acute withdrawal phase. Human and animal


models postulate that long-term use of opioids induces hypoadrenalism through impairment of the hypothalamic-pituitary-adrenal (HPA) axis. Opioid withdrawal leads to marked elevations of cortisol as a result of excess ACTH secretion (26, 32, 35). This HPA activation persists following normalization of the adrenergic system, which led some authors to conclude that cortisol is a more sensitive indicator of opioid withdrawal than catecholamines (30, 32). A small study by Higgins et al. on 5 non-dependent subjects assessed acute opioid withdrawal after a single dose of morphine and observed a dose-dependent increase in cortisol levels when subjects were subsequently injected with naloxone (28). Despite the clinical relevance, several limitations reduce the applicability of those results to our study population, mainly the selection of opioid-dependent subjects and rapid induction of withdrawal – through injection of naloxone or abrupt cessation of opioid with support medications such as alpha<sub>2</sub>-agonists. Since our subjects are mostly opioid-naive prior to hospitalization and will be gradually weaned off their opioids, the magnitude of increase in cortisol levels will likely be lower.

As for catecholamines, serum epinephrine and norepinephrine appear to increase rapidly following opioid withdrawal in numerous animal and human studies (12, 39-43). However, in contrast with cortisol, catecholamine levels decrease shortly following acute withdrawal. In a study of subjects undergoing rapid opioid detoxification, catecholamine levels peaked two hours following naloxone administration (12). A gradual opioid weaning as often seen in clinical practice is unlikely to be recognized through measurement of serum catecholamines.

# 3. Research objectives

#### Research question

What are the signs and symptoms of opioid-associated iatrogenic withdrawal syndrome (OIWS) in the adult ICU population?

#### Primary objective

To identify specific signs and symptoms of OIWS in mechanically ventilated adult ICU patients receiving at least 72 hours of regular opioids at the Montreal General Hospital (MGH) and the Royal Victoria Hospital (RVH) from February to October 2018

#### Secondary objective

To determine if the presence of OIWS is associated with an increase in serum cortisol.

#### 4. Methods

#### 4.1 Study design

### Multicenter Prospective Observational Open Cohort Study

The clinical presentation of OIWS is poorly described in the adult ICU population. The descriptive study design aims to identify signs and symptoms of OIWS in the prospect of developing a validated bedside screening tool. The prospective approach will enable collection of all relevant information while limiting missing data and assessing for potential confounding variables.

Throughout the study, investigators will be blinded to the diagnosis of OIWS to reduce evaluation bias and increase internal validity. Additionally, on one occasion for each patient, OIWS evaluation will be performed by two physicians, allowing for inter-rater reliability. This will ensure accurate OIWS diagnosis and reduce information bias. Following transfer to the ward, one additional data collection will be performed to optimize OIWS detection.

The study will be conducted in two hospitals of the McGill University Health Centre (MUHC) with different ICU populations, hereby increasing the external validity of the results. The MGH is a Level I trauma center, whereas the RVH treats surgical and medical patients. Furthermore, a multicentric approach will increase the sample size and the likelihood of describing the syndrome adequately.


### 4.2 Populations

## **Target population**

Mechanically ventilated adult ICU patients receiving continuous or regular intermittent opioids for more than 72 hours

### Source population

Mechanically ventilated adult ICU patients admitted to the MGH and the RVH from February to October 2018 receiving continuous or regular intermittent opioids for more than 72 hours and meeting the inclusion and none of the exclusion criteria of the study

### Study population

Mechanically ventilated adult ICU patients admitted to the MGH and the RVH from February to October 2018 receiving at least 72 hours of continuous or intermittent opioids, meeting the inclusion and none of the exclusion criteria and consenting to participate in the study

#### 4.3 Subject selection mode

#### 4.3.1 Inclusion criteria

- Patients 18 years of age or older
- Admitted to the RVH and MGH intensive care units from February to October 2018
- Patients requiring mechanical ventilation and receiving continuous or regular intermittent opioids for at least 72 hours (calculated from the hour of administration of the first opioid dose)
  - Recent prospective observational studies in the PICU and adult ICU populations have demonstrated that iatrogenic withdrawal symptoms may develop following 3-5 days of continuous opioid therapy (5, 8)
  - o Patient will be considered as receiving regular intermittent opioids if more than half of the scheduled "as-needed" doses within 24 hours were administered.
    - In the event that only prn narcotics are prescribed on a q1h prn or q2h prn basis, patients will be eligible if ≥ 4 prn doses are required per day.
- Weaning of at least 10% from previous stable opioid dose
  - A weaning episode is defined as a ≥ 10% decrease in the total stable opioid dose received over 4 hours for opioid infusions and over 12 hours for intermittent opioid administration (22)
  - According to our previous experience (i.e. WAAICUP-1), the weaning definition of ≥
     10% was chosen for practical reasons (8)

#### 4.3.2 Exclusion criteria

- Patient for whom consent cannot be obtained
- Patient and/or family unable to communicate in French or English
  - o May interfere with obtaining informed consent and OIWS assessment
- Patient who is deaf without appropriate hearing aid
  - Hearing impairment may interfere with patient communication and assessment of signs and symptoms
- Imminent and predictable death (< 72 hours) according to medical team
- Patients receiving opioids for the purposes of palliative care or prescribed by the palliative care team.
- Severe brain injury, defined as Glasgow Coma Scale (GCS) score of 8 or less at ICU admission
- Moderate brain injury, defined as GCS between 9 and 12, with elevated intracranial pressure (ICP > 20 mmHg) which requires ICP monitoring and osmotherapy
  - Major confounding factors for withdrawal syndrome by causing shivering, sympathetic drive and autonomic disorders
- Acute neurological condition (e.g. status epilepticus, encephalopathy, stroke)
  - Potential confounders of OIWS assessment


- If the acute neurological condition resolves within 72 hours, the patient may be included in the study
- Substance abuse prior to ICU admission
  - Chronic alcohol use defined as alcohol consumption of more than 2 drinks/day and/or more than 14 drinks/week for men and 9 drinks/week for women (44)
  - Chronic use of illicit drugs and amphetamines (except amphetamines taken for therapeutic purposes) defined as a consumption of at least 3 times per week
  - Chronic use of opioids (e.g. transdermal fentanyl, methadone, hydromorphone, etc.)
     defined as a consumption of at least 3 times per week
  - May induce withdrawal and confound OIWS assessment (45)
  - Chronic consumption of these substances will be confirmed by the patient, family, or medical chart
- Admission to the ICU with substance overdose or alcohol withdrawal syndrome.
- Readmission to the MGH or RVH ICU during the recruitment period (limit of one study entry per patient)
- Spinal cord injury above the lumbar region
  - o Sympathetic response to withdrawal absent depending on site/level of injury
  - Assessment tools not validated in these patients (DSM-5, RASS, CAM-ICU, CPOT)
- Opioid tolerance prior to ICU admission, defined as regular daily use of opioids for a chronic medical condition or continuous opioid administration for > 7 days prior to ICU admission (46) Does not include patients who take opioids infrequently.
  - The FDA defines opioid tolerance as patients receiving at least 60 mg/day of oral morphine equivalents (600 mcg IV fentanyl IV equivalents/day) for ≥ 1 week (46)

#### 4.4 Definition of variables

### 4.4.1 Primary outcome variables

# Dependent variables

- Presence of signs and symptoms of OIWS
  - According to daily evaluation by investigator after an episode of opioid weaning has begun (See Appendix III)

#### Independent variables

- **Presence of OIWS** (qualitative nominal dichotomous)
  - According to DSM-5 evaluation completed daily by physician after an episode of opioid weaning has begun
- Demographic and clinical variables
  - o **Age** (quantitative continuous): Age in years at ICU admission
  - Sex (qualitative nominal dichotomous)
  - o **Weight** (quantitative continuous): Weight in kg at ICU admission
  - o **Height** (quantitative continuous): Height in cm at ICU admission
  - o **Body mass index** (BMI) (quantitative continuous): In kg/m<sup>2</sup> at ICU admission
  - Ethnicity (qualitative nominal)
  - o Site of ICU admission (qualitative nominal dichotomous)
  - Smoking status (qualitative nominal dichotomous)
    - Number of cigarettes per day according to medical chart, patient or family at ICU admission (quantitative discrete)
    - Number of pack-years according to medical chart, patient or family at ICU admission (quantitative continuous)
  - o Principal diagnosis at ICU admission (qualitative nominal)
    - Definite diagnosis according to medical chart at ICU admission using ICD-10 classification
  - Length of stay in the ICU (quantitative continuous)
    - Time in hours from ICU admission to ICU discharge, transfer to ward or patient death, according to medical chart
    - Opioid withdrawal has been associated with longer ICU stays (4-6)
  - Duration of mechanical ventilation (quantitative continuous)

- Time in hours according to medical chart
- Longer duration of mechanical ventilation has been associated with increased risk of IWS in ICU patients (7)
- Acute Physiology and Chronic Health Evaluation II Score (APACHE II) (qualitative ordinal)
  - To assess severity of disease and ICU mortality on a scale of 0 to 71 (47)
  - As reported by an archivist based on data from the first 24 hours of ICU admission
- Glasgow Coma Scale (GCS) (qualitative ordinal)
  - To assess mental status and severity of brain injury on a scale of 3 to 15 (48)
  - As reported by nurse on patient flow sheet at ICU admission

#### **Renal function**

- Daily serum creatinine in umol/L according to medical chart (quantitative continuous)
- Presence of renal replacement therapy according to medical chart (qualitative nominal - dichotomous)
- Drug accumulation may occur when renal excretion is decreased, minimizing **OIWS**

#### Level of hepatic dysfunction upon ICU admission

- Severity of hepatic dysfunction as calculated by the Child-Turcotte-Pugh score at ICU admission (qualitative ordinal)
- Drug accumulation may occur when hepatic metabolism is decreased
- **Presence of ECMO** (qualitative nominal dichotomous)
  - Collected daily according to medical chart
  - Patients on ECMO may require higher fentanyl doses due to sequestration of lipophilic drugs and increased volume of distribution (49)
- **Cumulative opioid dose preweaning** (quantitative continuous)
  - Cumulative opioid dose in fentanyl equivalents (µg/kg) according to medication administration record (MAR) from time of start of opioids during ICU admission
  - Higher cumulative opioid doses have been associated with increased risk of IWS in ICU patients (8)
- **Duration of continuous opioid administration preweaning** (quantitative continuous)
  - Time in hours according to MAR or patient flow sheet
  - Prolonged opioid exposure has been associated with an increased risk of IWS in ICU patients (4, 8, 13-15)
- Rate of opioid weaning > 10% from previous stable dose (quantitative continuous)
  - Calculated in % according to MAR or patient flow sheet
    - Continuous infusion: perfusion rate over previous 4h
      - Continuous intermittent administration: total dose over previous 12h
  - Rapid tapering or abrupt discontinuation of opioids has been associated with increased risk of IWS in ICU patients (7, 20)
- Presence of clonidine, beta-blockers or antidepressants prior to ICU admission (aualitative nominal - dichotomous)
  - The agent and whether it was represcribed in ICU will be noted according to the medication reconciliation chart at admission
  - These medications may cause withdrawal when discontinued
- Occasional use of prescribed opioids prior to ICU admission (qualitative nominal dichotomous)
  - Agent (qualitative nominal) and daily doses in fentanyl equivalents (µg/kg/day) (quantitative continuous) will be noted according to medication reconciliation chart at admission
  - Chronic opioid users are excluded from the present study (as indicated in exclusion criteria)

- **Prior history of substance abuse** (qualitative nominal dichotomous)
  - Agent (qualitative nominal) will be noted according to patient, family or medical chart
  - A prior history of substance abuse may render those patients more susceptible to CNS depressants (e.g. opioids and benzodiazepines)

#### Confounding variables

- Chronic or occasional use of benzodiazepines prior to ICU admission (qualitative nominal dichotomous)
  - Agent (qualitative nominal) and total daily doses in lorazepam equivalents (mg/kg/day) (quantitative continuous) will be noted according to medication reconciliation chart at admission
  - Withdrawal due to benzodiazepines may overlap with OIWS assessment (6, 24)
- Concomitant administration of benzodiazepines during ICU stay (qualitative nominal dichotomous)
  - Agent and total daily dose (mg/kg) will be noted daily (qualitative nominal and quantitative continuous, respectively), as well as total cumulative benzodiazepine dose received since ICU admission in lorazepam equivalents (mg/kg) (quantitative continuous), according to MAR.
  - Higher mean daily doses of benzodiazepines have been associated with an increased risk of IWS in ICU patients (7)
  - Withdrawal due to benzodiazepines may overlap with OIWS assessment (6, 24)
- Administration of medication that may influence severity of OIWS (e.g. clonidine, dexmedetomidine, methadone, buprenorphine, propofol, beta-blockers and antipsychotics) (qualitative nominal - dichotomous)
  - Agent, total daily dose will be noted daily according to MAR (qualitative nominal)
  - Clonidine, dexmedetomidine, methadone, buprenorphine and antipsychotics can be used to treat or attenuate symptoms of opioid withdrawal and therefore may confound OIWS assessment (4, 50)
- Presence of chronic neurological conditions (e.g. dementia, Parkinson's disease, essential tremor) (qualitative nominal - dichotomous)
  - According to past medical history in medical chart
  - Symptoms of dementia and Parkinson's disease may confound OIWS assessment
- **Presence of delirium** (qualitative nominal dichotomous)
  - During ICU stay: according to the Confusion Assessment Method for the ICU (CAM-ICU) as measured by investigators during evaluation and/or nursing staff, collected daily once opioid weaning is initiated and until transfer
  - After transfer to ward: according to the Confusion Assessment Method (CAM) measured once by investigators within 24-96 hours of transfer
  - Symptoms of delirium may overlap with OIWS assessment (10, 20, 51)
- Presence of agitation due to a condition other than OIWS (qualitative nominal dichotomous) (10)
  - During ICU stay: according to the Richmond Agitation-Sedation Scale (RASS) as measured by investigators and/or nursing staff, collected daily once opioid weaning is initiated (auglitative ordinal) and until transfer
  - After transfer to ward: according to the Agitated Behavior Scale (ABS), measured once by investigators within 24-96 hours of transfer (qualitative ordinal)
- **Presence of pain** (qualitative nominal dichotomous)
  - In patients unable to self-report: Critical-Care Pain Observation Tool (CPOT) score > 2, as measured by investigator or medical staff, collected daily once opioid weaning is initiated
  - In patients able to self-report: Numeric Rating Scale (NRS) ≥ 4, collected daily once opioid weaning is initiated
  - The symptoms of uncontrolled pain may confound OIWS assessment (20)

- Administration of co-analgesia during ICU hospitalization (e.g. acetaminophen, non-steroidal anti-inflammatory drugs, anticonvulsants, antidepressants, corticosteroids) (qualitative nominal)
  - Agent and total daily dose will be noted daily according to MAR
  - Co-analgesia is used to treat or attenuate pain, which may confound OIWS assessment
  - Anti-inflammatory drugs also act as antipyretics, which may confound OIWS assessment
- **Presence of nicotine replacement therapy during ICU admission** (qualitative nominal dichotomous)
  - Nicotine consumption in mg (qualitative continuous) prior to ICU admission (e.g. cigarettes, nicotine replacement therapy) and whether nicotine replacement therapy was prescribed in ICU will be noted according to medication reconciliation chart at admission (qualitative nominal)
  - Nicotine withdrawal or nicotine-induced delirium may confound OIWS assessment (45)
- Factors which may confound specific signs and symptoms of OIWS (qualitative nominal dichotomous)
  - Fever secondary to documented or suspected infection
    - According to diagnosis documented in medical chart
  - Diarrhea due to Clostridium difficile infection or enteral feeds
    - According to positive C. difficile antigen detection test in medical chart or presence of enteral feeds in patient flow sheet
- **Use of physical restraints** (qualitative nominal dichotomous) (52)
  - Collected daily according to medical chart
  - Patients with restraints are more likely to be given supplemental sedative and analgesic agents which may confound OIWS assessment

### 4.4.2 Secondary outcome variables

Both serum cortisol levels will only be measured in patients not receiving exogenous corticosteroids.

#### Independent variables

- **Basal serum cortisol level** (quantitative continuous)
  - Measured ± 2 hours from the start of opioid weaning
- **Weaning serum cortisol level** (quantitative continuous)
  - Measured on the day of transfer to ward or after a maximum of 72 hours after start of weaning, at the same time of day as the first measure, whichever occurs first.
- Change in serum cortisol levels (quantitative continuous)
  - Difference between weaning and basal serum cortisol levels

## **Confounding variables**

- **Timing of sample in hh:mm** (quantitative continuous)
  - Cortisol is secreted in a diurnal pattern (53)
  - Serum cortisol samples will be taken at the same time of day
- Presence of primary adrenal insufficiency (qualitative nominal dichotomous)
  - According to past medical history in medical chart
  - Patients with this condition may present with hypocortisolemia and receive exogenous corticosteroids, which may confound serum cortisol assays
- Presence of acute illness (infection, trauma, surgery, illness) (qualitative nominal)
  - According to APACHE II score at ICU admission
  - Cortisol has been studied as a marker of severity of disease, with higher levels associated with worse prognosis. This association appears to be stronger during the first two days of admission (54)
  - May thus increase cortisol levels depending on severity of disease (53)

- May also provoke transient adrenal insufficiency (53)
- Presence of septicemia or septic shock (qualitative nominal dichotomous)
  - Diagnosis of sepsis will be noted according to medical chart
  - Sepsis causes relative adrenal insufficiency in up to 30 to 70% of patients, which may confound results (55-57)
- Medications (ketoconazole, spironolactone, dopamine agonists, etc.) (qualitative nominal)
  - May reduce cortisol production (53)

# 4.5 Data collection and study procedure (Appendix II)

From February to October 2018, patients from the MGH and RVH critical care units will be screened daily from unit patient lists generated through Oasis for eligibility. The investigators will be transiting daily between both centers. Once a patient is approaching 72 hours of mechanical ventilation and regular opioid administration, subjects will be evaluated for inclusion and exclusion criteria according to medical chart, and data will be recorded in the "Patient Screen Log". Once a patient fits our entry criteria, here are the steps for obtaining consent:

- 1- A member of the treating team (ICU physician or patient nurse) will inform the patient about this research project. If the patient is deemed unfit to provide informed consent, the patient's decision maker will be approached.
- 2- If patient/decision maker shows interest, a member of the research team, independent of the clinical care of the patient will meet with the patient/decision maker and explain the research and seek informed consent.
- 3- If the intubated patient verbally agrees but is unable to sign the consent, then a witness will sign the consent and the discussion will be documented on the consent form.
- 4- If the consent is obtained from a decision maker, then we will further seek direct patient consent as soon as patient is deemed apt to consent.

In this case, we would ask the patient to sign a new consent form and a copy will be provided to the patient and the newly signed consent will be kept in our files.

Once recruitment is completed, the patient will be given a subject number and placed on the "Enrollment List", which includes medical record numbers, admission dates, screen dates and enrollment dates.

After enrollment, demographic, reason for admission, lifestyle and medical data will be collected retrospectively from the medical chart, the patient's family and the medical team, and will be noted in the "Enrollment and Outcomes Form". The reasons for exclusion and the number of patients who refused consent will be collected. Temporarily excluded patients will be re-evaluated daily for possible inclusion into the study.

Once the patient begins the targeted opioid weaning of  $\geq$  10%, investigators will perform evaluations daily between 10am and 2pm. These evaluations will consist of using pre-tested data collection sheets to record signs and symptoms of possible OIWS, opioid doses, administered medications, laboratory values and other clinical data such as the RASS, CPOT and CAM-ICU scores. Data collection will be based on subject observation and interview when possible, nurse assessments, medical charts and laboratory results. Serum cortisol levels will be measured on the first day of opioid weaning ( $\pm$  2 hours from dose decrease) and on the day patient is transferred to the ward or 72 hours from start of weaning whichever occurs first.

Once a weaning episode is identified, the physician collaborator will be contacted to perform daily DSM-5 evaluations. DSM-5 evaluations will be placed in opaque envelopes and investigators will be blinded to the results throughout the study. Additionally, for each patient, at least one inter-rater DSM-5 evaluation between 2 physician collaborators will be performed in order to assess interrater reliability. The two evaluations will be done within 2 hours of each other to minimize time-related discrepancies.


If opioid weaning is unsuccessful and opioid dose is re-increased, the subject will continue to be observed, however daily evaluations will only resume at the next weaning episode. Daily follow-up ends on day of transfer to the ward. One additional data collection and DSM-5 evaluation will be performed on the same day within 24 to 96 hours following transfer. Follow up ends 14 days after initial opioid weaning if patient remains in the ICU or if patient dies.

### 4.6 Measurement tools

| DSM-5<br>(Appendix IV) | <ul> <li>No validated diagnostic tools for OIWS currently exist in the adult ICU</li> <li>DSM-5 is the gold standard for diagnosing opioid withdrawal in numerous settings</li> <li>Although not validated in the ICU population, it remains the most appropriate OIWS diagnostic tool for the study (9, 58)</li> </ul> |
|---|---|
| APACHE II score<br>(Appendix V) | <ul> <li>Validated tool to predict the risk of mortality in ICU patients (47, 59)</li> <li>Calculated by an archivist using data collected in the first 24h of ICU admission</li> <li>In this study: to assess patient disease severity at enrollment</li> </ul> |
| Glasgow Coma<br>Scale (GCS)<br>(Appendix VI) | <ul> <li>Validated in ICU and trauma patients to assess the severity of head trauma based on ocular, verbal and motor criteria (48)</li> <li>GCS score ≤ 8: comatose patient with no evidence of eye or verbal response</li> <li>GCS score 9-15: presence of eye and verbal response (60)</li> <li>In this study: to assess the level of consciousness of trauma patients and to verify exclusion criteria at ICU admission</li> </ul> |
| Child-Turcotte-<br>Pugh score<br>(Appendix VII) | <ul> <li>Extensively studied in critically ill patients to assess liver function (61)</li> <li>In the ICU, CTP scores at admission correlate with 12-month mortality (62)</li> <li>In this study: to assess severity of hepatic dysfunction at ICU admission</li> </ul> |
| Confusion Assessment Method (CAM) (Appendix IX) | <ul> <li>Validated tool to identify delirium in patients on general medicine hospital wards</li> <li>Enables non-psychiatrist clinicians to quickly determine if delirium is present (63)</li> <li>In this study: performed by the investigator within 24-96 hours of ICU transfer to ward</li> </ul> |
| CAM-ICU<br>(Appendix VIII) | - Validated tool to identify presence of delirium in a dichotomous manner in the ICU (64) - In this study: collected daily by investigators or according to nurse assessment |
| Richmond<br>Agitation<br>Assessment<br>Scale (RASS)<br>(Appendix X) | <ul> <li>To assess level of agitation and sedation, and to prevent under or over sedation in ICU</li> <li>Scale ranges from -5 (unarousable sedation) to +4 (combative)</li> <li>RASS score ≤ -3 indicates a deeply sedated state (65)</li> <li>In this study: collected daily by investigator and according to nurse assessment</li> <li>RASS + 1 defines restlessness and RASS ≥ 2 defines agitation</li> </ul> |
| Agitated Behaviour Scale (ABS) (Appendix XI) | <ul> <li>Originally designed to assess agitation in patients with traumatic brain injury (66)</li> <li>Validated in numerous settings, including long-term care facility (67)</li> <li>ABS score ≥ 22: Agitation, ≤ 21: No agitation (68)</li> <li>In this study: performed once by the investigator within 24-96h of ICU transfer</li> </ul> |
| Critical-Care Pain Observation Tool (CPOT) (Appendix XII) | <ul> <li>To assess pain in critically ill mechanically ventilated patients based on facial expressions, body movements and muscle tension during nociceptive procedures</li> <li>To qualify pain in patients unable to verbalize; in patients able to communicate, self-reporting of pain remains the gold standard</li> <li>CPOT &gt; 2: unacceptably high level of pain, ≤ 2: minimal to no pain (68)</li> <li>In this study: measured daily by investigators and according to nurse assessment</li> </ul> |
| Numeric Rating | - To assess pain intensity on a numerical scale, most commonly ranging from 0 to 10 |


# Scale (NRS) (Appendix XIII)

(NRS-11); only the scale extremities are detailed (69)

- In this study: to assess pain during daily evaluations once patients can self-report. Investigators will ask patients to rate their pain on a scale from 0 (absence of pain) to 10 (worst pain imaginable). An NRS  $\geq$  4 represents an unacceptable level of pain.

#### 5. Data analysis

# 5.1 Statistical analysis

## 5.1.1 Descriptive statistics

Demographic and clinical characteristics of patients who developed OIWS will be compared to those who did not. Categorical variables will be presented as proportions. For continuous variables, means and standard deviations will be computed for normal distributions whereas medians (interquartile range) will be used for non-normal distributions.

For the primary outcome, episodes will be compared between the withdrawal positive (W+) group and the withdrawal negative (W-) group. Every day on which the DSM-5 is positive is equivalent to an episode of withdrawal, whereas a negative DSM-5 counts as an episode in which no withdrawal was observed. Patients who are positive for at least one episode of withdrawal make up the W+ group, whereas those who did not have a single episode of withdrawal make up the W- group, thus eliminating crossover. If a single patient experiences multiple days of withdrawal, s/he will account for multiple episodes in the study. Signs and symptoms will be tallied per episode and compared between the two groups. The results will be presented as proportions (i.e. incidence of symptom per total episodes). In the event of a discordant inter-rater evaluation, only the positive result will be taken into account.

For the secondary outcome, serum cortisol levels and changes in serum cortisol levels are continuous variables and therefore descriptive statistics will be used as stated above, depending on the distribution.

#### 5.1.2 Statistical inference

To gauge for presence of evaluation bias, inter-rater agreement will be determined using Cohen's kappa. This test measures the extent to which physicians concur when assessing for presence of OIWS using the DSM-5 criteria. A kappa of  $\geq$  0.61 is indicative of good inter-rater agreement (70).

For secondary outcomes, baseline, weaning and change in cortisol levels will be compared between patients positive and negative for OIWS. A Student's t-test or a Wilcoxon signed rank test will be used. The test will be determined based on distribution and sample size.

#### 5.2 Sample size

Based on our experience with the WAAICUP studies, 88 patients were eligible to participate in the study in an 8-month period, of which around 50 consented (22). We thus aim to recruit 50 patients based on the feasibility of these previous studies.

#### 6. Advantages and limitations

## 6.1 Advantages

As stated previously, a prospective approach will limit missing data and enable assessment of potential confounders. The multicentric design enables study of different ICU populations, thereby increasing external validity and sample size.

There is currently no validated tool for OIWS diagnosis in the adult ICU population. Use of the DSM-5 is adequate in this study since it standardizes physician evaluation and is considered a gold standard in numerous settings. Multiple other ICU-validated tools will be used throughout the study such as the RASS, CAM-ICU and CPOT. Validated tools will also be used after transfer to the ward.


Training will be provided to investigators in order to standardize assessment and reduce observer bias. Observer bias will also be minimized by the blinding of investigators to DSM-5 results. Additionally, DSM-5 inter-rater agreement will be assessed on one occasion for each patient. A notable advantage is the supplemental follow-up after transfer to ward, which increases internal validity by limiting loss of patients who might develop OIWS later once transferred out of the ICU.

To our knowledge, no previous study has explored potential biomarkers that correlate with symptoms of OIWS. The exploratory use of serum cortisol in this study is thus a novel research avenue and will enable further characterization of OIWS.

#### **6.2 Limitations**

The study is susceptible to several limitations, most of them due to study design Due to lack of randomization, the study is subject to confounding. A notable covariate is the concomitant administration of benzodiazepines, which is difficult to control for since ICU patients frequently receive both opioids and benzodiazepines, and there is significant overlap in their respective withdrawal symptoms. However, administration of benzodiazepines will be noted during daily evaluations. The study is also susceptible to the "clinical trial effect" bias, since the attending physicians are not blinded to patient enrollment in the study and may modify their management consequently. To control for observer bias, pre-tested standardized data collection forms will be used, but it does not eliminate it completely, as evaluations will be performed by different investigators.

Since the sample size was determined on the basis of feasibility rather than statistical power, no statistically significant associations can be made. Statistical analyses will thus be predominantly descriptive in nature.

The exclusion of patients with severe or moderate traumatic brain injury requiring ICP monitoring and osmotherapy reduces external validity. These patients are important consumers of opioids and are therefore at risk of developing OIWS. However, their clinical condition would make the adequate assessment of OIWS impossible.

#### 7. Relevance of study

To our knowledge, this is the first prospective study that aims to describe the clinical presentation of OIWS in the adult ICU setting with a standardized approach, fulfilling an identified research gap (71). As mentioned, OIWS is a clinical entity associated with negative outcomes that is poorly understood in critically ill adults because of diagnostic challenges. With a more accurate description of the clinical presentation, it would be possible to develop reliable screening tools to identify patients most at risk of OIWS and to sensitize the clinician to adopt appropriate measures in their management. An accurate description of the clinical presentation of OIWS is the first step in a series of research advances aimed at correctly recognizing and managing OIWS in adult ICU patients.

### 8. Ethical considerations and patient consent

The study protocol will be approved by the MUHC Research Ethics Board prior to enrollment. The study procedure does not require direct medical intervention as it is observational in design. The evaluation of signs and symptoms will mostly be done using ICU standard of care assessment tools (e.g. CAM-ICU, CPOT, RASS). Assessments that are not part of routine ICU care include collection of two blood samples per patient for serum cortisol measurement and DSM-5. Investigators will not interfere with usual care, which prevents patient exposure to additional risk

Written and informed consent will be obtained prior to enrollment and a copy will be given to the patient. Consent forms will be available in English and French with detailed descriptions of the study procedure and interventions. If the patient is inapt, consent will be obtained from a legal representative (e.g. family member). Once the patient is apt, direct consent will be sought. If the


patient refuses consent, previously collected data will be destroyed. Patients or their legal representative may decide to withdraw from the study at any moment.

Patient confidentiality will be maintained throughout the study by various means. All data will be deidentified and coded. The code will be maintained by the principle investigator. Computers and files will be password protected. Paper data will be kept in opaque envelopes in a locked cabinet to which only the investigators will have access. Study data will be kept for 7 years and the study itself will be registered on clinicaltrials.gov.


#### 9. References

- 1. Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, et al. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013;41(1):263-306.
- 2. Burry LD, Williamson DR, Perreault MM, Rose L, Cook DJ, Ferguson ND, et al. Analgesic, sedative, antipsychotic, and neuromuscular blocker use in Canadian intensive care units: a prospective, multicentre, observational study. Canadian Journal of Anesthesia/Journal canadien d'anesthésie. 2014;61(7):619-30.
- 3. Best KMPRN, Wypij DP, Asaro LAMS, Curley MAQPRNF, for the Randomized Evaluation of Sedation Titration For Respiratory Failure Study I. Patient, Process, and System Predictors of latrogenic Withdrawal Syndrome in Critically III Children\*. Critical Care Medicine. 2017;45(1):e7-e15.
- 4. Chiu AW, Contreras S, Mehta S, Korman J, Perreault MM, Williamson DR, et al. latrogenic Opioid Withdrawal in Critically III Patients: A Review of Assessment Tools and Management. Ann Pharmacother. 2017;51(12):1099-111.
- 5. da Silva PS, Reis ME, Fonseca TS, Fonseca MC. Opioid and Benzodiazepine Withdrawal Syndrome in PICU Patients: Which Risk Factors Matter? J Addict Med. 2016;10(2):110-6.
- 6. Amigoni A, Mondardini MC, Vittadello I, Zaglia F, Rossetti E, Vitale F, et al. Withdrawal Assessment Tool-1 Monitoring in PICU: A Multicenter Study on latrogenic Withdrawal Syndrome. Pediatric Critical Care Medicine. 2017;18(2):e86-e91.
- 7. Cammarano WB, Pittet JF, Weitz S, Schlobohm RM, Marks JD. Acute withdrawal syndrome related to the administration of analgesic and sedative medications in adult intensive care unit patients. Crit Care Med. 1998;26(4):676-84.
- 8. Wang PP, Huang E, Feng X, Bray C-A, Perreault MM, Rico P, et al. Opioid-associated iatrogenic withdrawal in critically ill adult patients: a multicenter prospective observational study. Annals of Intensive Care. 2017;7(1):88.
- 9. Duceppe MA, Perreault MM, Frenette AJ, Burry L, Rico L, Lavoie A, et al. latrogenic withdrawal from opioids and benzodiazepines in the intensive care unit: a systematic review. Submitted to Crit Care Medicine Dec 2017.
- 10. Harris J, Ramelet AS, van Dijk M, Pokorna P, Wielenga J, Tume L, et al. Clinical recommendations for pain, sedation, withdrawal and delirium assessment in critically ill infants and children: an ESPNIC position statement for healthcare professionals. Intensive Care Med. 2016;42(6):972-86.
- 11. Anand KJ, Willson DF, Berger J, Harrison R, Meert KL, Zimmerman J, et al. Tolerance and withdrawal from prolonged opioid use in critically ill children. Pediatrics. 2010;125(5):e1208-25.
- 12. Gerra G, Ceresini S, Esposito A, Zaimovic A, Moi G, Bussandri M, et al. Neuroendocrine and behavioural responses to opioid receptor-antagonist during heroin detoxification: relationship with personality traits. Int Clin Psychopharmacol. 2003;18(5):261-9.
- 13. Brown C, Albrecht R, Pettit H, McFadden T, Schermer C. Opioid and benzodiazepine withdrawal syndrome in adult burn patients. Am Surg. 2000;66(4):367-70; discussion 70-1.
- 14. Dominguez KD, Lomako DM, Katz RW, Kelly HW. Opioid withdrawal in critically ill neonates. Ann Pharmacother. 2003;37(4):473-7.
- 15. Ista E, de Hoog M, Tibboel D, Duivenvoorden HJ, van Dijk M. Psychometric evaluation of the Sophia Observation withdrawal symptoms scale in critically ill children. Pediatr Crit Care Med. 2013;14(8):761-9.
- 16. Best KM, Boullata JI, Curley MA. Risk factors associated with iatrogenic opioid and benzodiazepine withdrawal in critically ill pediatric patients: a systematic review and conceptual model. Pediatric critical care medicine: a journal of the Society of Critical Care Medicine and the World Federation of Pediatric Intensive and Critical Care Societies. 2015;16(2):175-83.
- 17. Fisher D, Grap MJ, Younger JB, Ameringer S, Elswick RK. Opioid withdrawal signs and symptoms in children: frequency and determinants. Heart Lung. 2013;42(6):407-13.
- 18. Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, et al. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002;30(1):119-41.


- 19. Ista E, van Dijk M, de Hoog M, Tibboel D, Duivenvoorden HJ. Construction of the Sophia Observation withdrawal Symptoms-scale (SOS) for critically ill children. Intensive Care Med. 2009;35(6):1075-81.
- 20. Ista E, van Dijk M, Gamel C, Tibboel D, de Hoog M. Withdrawal symptoms in critically ill children after long-term administration of sedatives and/or analgesics: a first evaluation. Crit Care Med. 2008;36(8):2427-32.
- 21. Franck LS, Naughton I, Winter I. Opioid and benzodiazepine withdrawal symptoms in paediatric intensive care patients. Intensive Crit Care Nurs. 2004;20(6):344-51.
- 22. Perreault MM MA, Sandu PR, Rosu VA, Capilnean A, Murgoi P, et al., editor Withdrawal assessment in adult ICU patients: validation of the WAT-1 scale. 37th International Symposium on Intensive Care and Emergency Medicine; 2017.
- 23. Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003;35(2):253-9.
- 24. Ista E, van Dijk M, Gamel C, Tibboel D, de Hoog M. Withdrawal symptoms in children after long-term administration of sedatives and/or analgesics: a literature review. "Assessment remains troublesome". Intensive Care Med. 2007;33(8):1396-406.
- 25. Barr MC, Huitron-Resendiz S, Sanchez-Alavez M, Henriksen SJ, Phillips TR. Escalating morphine exposures followed by withdrawal in feline immunodeficiency virus-infected cats: a model for HIV infection in chronic opiate abusers. Drug Alcohol Depend. 2003;72(2):141-9.
- 26. Cami J, Gilabert M, San L, de la Torre R. Hypercortisolism after opioid discontinuation in rapid detoxification of heroin addicts. Br J Addict. 1992;87(8):1145-51.
- 27. Elman I, D'Ambra MN, Krause S, Breiter H, Kane M, Morris R, et al. Ultrarapid opioid detoxification: effects on cardiopulmonary physiology, stress hormones and clinical outcomes. Drug Alcohol Depend. 2001;61(2):163-72.
- 28. Higgins ST, Preston KL, Cone EJ, Henningfield JE, Jaffe JH. Supersensitivity to naloxone following acute morphine pretreatment in humans: behavioral, hormonal and physiological effects. Drug Alcohol Depend. 1992;30(1):13-26.
- 29. Wen HL, Ho WK, Wong HK, Mehal ZD, Ng YH, Ma L. Changes in adrenocorticotropic hormone (ACTH) and cortisol levels in drug addicts treated by a new and rapid detoxification procedure using acupuncture and naloxone. Comp Med East West. 1979;6(3):241-5.
- 30. Culpepper-Morgan JA, Kreek MJ. Hypothalamic-pituitary-adrenal axis hypersensitivity to naloxone in opioid dependence: a case of naloxone-induced withdrawal. Metabolism. 1997;46(2):130-4.
- 31. Hellman L, Fukushima DK, Roffwarg H, Fishman J. Changes in estradiol and cortisol production rates in men under the influence of narcotics. J Clin Endocrinol Metab. 1975;41(06):1014-9.
- 32. Nava F, Caldiroli E, Premi S, Lucchini A. Relationship between plasma cortisol levels, withdrawal symptoms and craving in abstinent and treated heroin addicts. J Addict Dis. 2006;25(2):9-16.
- 33. Shi J, Li SX, Zhang XL, Wang X, Le Foll B, Zhang XY, et al. Time-dependent neuroendocrine alterations and drug craving during the first month of abstinence in heroin addicts. Am J Drug Alcohol Abuse. 2009;35(5):267-72.
- 34. Vargas ML, Gonzalvez ML, Martinez JA, Arias L, Bruger AJ, Milanes MV. Effects of clonidine on pituitary-adrenocortical axis in morphine-tolerant rats and after naloxone-induced withdrawal. Pharmacology. 1992;44(3):158-64.
- 35. Zhang GF, Ren YP, Sheng LX, Chi Y, Du WJ, Guo S, et al. Dysfunction of the hypothalamic-pituitary-adrenal axis in opioid dependent subjects: effects of acute and protracted abstinence. Am J Drug Alcohol Abuse. 2008;34(6):760-8.
- 36. Cachat J, Canavello P, Elegante M, Bartels B, Hart P, Bergner C, et al. Modeling withdrawal syndrome in zebrafish. Behav Brain Res. 2010;208(2):371-6.
- 37. Bearn J, Buntwal N, Papadopoulos A, Checkley S. Salivary cortisol during opiate dependence and withdrawal. Addict Biol. 2001;6(2):157-62.
- 38. Rabbani M, Hajhashemi V, Mesripour A. Increase in brain corticosterone concentration and recognition memory impairment following morphine withdrawal in mice. Stress (Amsterdam, Netherlands). 2009;12(5):451-6.


- 39. Brent PJ, Johnston PA, Chahl LA. Plasma catecholamine concentrations during morphine withdrawal in conscious guinea-pigs. Clin Exp Pharmacol Physiol. 1987;14(8):623-31.
- 40. Chang AP, Dixon WR. Role of plasma catecholamines in eliciting cardiovascular changes seen during naloxone-precipitated withdrawal in conscious, unrestrained morphine-dependent rats. J Pharmacol Exp Ther. 1990;254(3):857-63.
- 41. Weil-Malherbe H, Smith ER, Eisenman AJ, Fraser HF. Plasma catecholamine levels and urinary excretion of catecholamines and metabolites in two human subjects during a cycle of morphine addiction and withdrawal. Biochem Pharmacol. 1965;14(11):1621-33.
- 42. Delle M, Ricksten SE, Haggendal J, Olsson K, Skarphedinsson JO, Thoren P. Regional changes in sympathetic nerve activity and baroreceptor reflex function and arterial plasma levels of catecholamines, renin and vasopressin during naloxone-precipitated morphine withdrawal in rats. J Pharmacol Exp Ther. 1990;253(2):646-54.
- 43. McDonald T, Hoffman WE, Berkowitz R, Cunningham F, Cooke B. Heart rate variability and plasma catecholamines in patients during opioid detoxification. J Neurosurg Anesthesiol. 1999;11(3):195-9.
- 44. Québec INdSPd. Public Policy and Health. Alcohol Consumption and Public Health in Québec : Summary: Gouvernement du Québec ; 2013.
- 45. Awissi DK, Lebrun G, Fagnan M, Skrobik Y, Regroupement de Soins Critiques RdSRQ. Alcohol, nicotine, and iatrogenic withdrawals in the ICU. Crit Care Med. 2013;41(9 Suppl 1):S57-68.
- 46. Administration USFaD. EXTENDED-RELEASE (ER) AND LONG-ACTING (LA) OPIOID ANALGESICS RISK EVALUATION AND MITIGATION STRATEGY (REMS). 2015.
- 47. Capuzzo M, Valpondi V, Sgarbi A, Bortolazzi S, Pavoni V, Gilli G, et al. Validation of severity scoring systems SAPS II and APACHE II in a single-center population. Intensive Care Med. 2000;26(12):1779-85.
- 48. Moore L, Lavoie A, Camden S, Le Sage N, Sampalis JS, Bergeron E, et al. Statistical validation of the Glasgow Coma Score. J Trauma. 2006;60(6):1238-43; discussion 43-4.
- 49. Marhong JD, DeBacker J, Viau-Lapointe J, Munshi L, Del Sorbo L, Burry L, et al. Sedation and Mobilization During Venovenous Extracorporeal Membrane Oxygenation for Acute Respiratory Failure: An International Survey. Crit Care Med. 2017;45(11):1893-9.
- 50. Prunty JM, J. PJ. Acute Opioid Withdrawal Identification and Treatment Strategies. [EPub]2016.
- 51. Devlin JW, Mallow-Corbett S, Riker RR. Adverse drug events associated with the use of analgesics, sedatives, and antipsychotics in the intensive care unit. Crit Care Med. 2010;38(6 Suppl):\$231-43.
- 52. Lucidarme O, Seguin A, Daubin C, Ramakers M, Terzi N, Beck P, et al. Nicotine withdrawal and agitation in ventilated critically ill patients. Crit Care. 2010;14(2):R58.
- 53. Cooper MS, Stewart PM. Corticosteroid insufficiency in acutely ill patients. N Engl J Med. 2003;348(8):727-34.
- 54. Tarjanyi Z, Montsko G, Kenyeres P, Marton Z, Hagendorn R, Gulyas E, et al. Free and total cortisol levels are useful prognostic markers in critically ill patients: a prospective observational study. Eur J Endocrinol. 2014;171(6):751-9.
- 55. Dubey A, Boujoukos AJ. Measurements of serum free cortisol in critically ill patients. Crit Care. 2004;9(1):E2.
- 56. Annane D, Briegel J, Sprung CL. Corticosteroid insufficiency in acutely ill patients. N Engl J Med. 2003;348(21):2157-9.
- 57. Annane D, Maxime V, Ibrahim F, Alvarez JC, Abe E, Boudou P. Diagnosis of adrenal insufficiency in severe sepsis and septic shock. Am J Respir Crit Care Med. 2006;174(12):1319-26.
- 58. APA. Diagnostic and Statistical Manual of Mental Disorders: DSM-5. American Psychiatric Publishing. 5th ed. ed. Washington, DC2013.
- 59. Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985;13(10):818-29.
- 60. Teasdale G, Jennett B, Murray L, Murray G. Glasgow coma scale: to sum or not to sum. Lancet. 1983;2(8351):678.


- 61. Saliba F, Ichai P, Levesque E, Samuel D. Cirrhotic patients in the ICU: prognostic markers and outcome. Curr Opin Crit Care. 2013;19(2):154-60.
- 62. Warren A, Soulsby CR, Puxty A, Campbell J, Shaw M, Quasim T, et al. Long-term outcome of patients with liver cirrhosis admitted to a general intensive care unit. Ann Intensive Care. 2017;7(1):37.
- 63. Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008;56(5):823-30.
- 64. Gusmao-Flores D, Salluh JI, Chalhub RA, Quarantini LC. The confusion assessment method for the intensive care unit (CAM-ICU) and intensive care delirium screening checklist (ICDSC) for the diagnosis of delirium: a systematic review and meta-analysis of clinical studies. Crit Care. 2012;16(4):R115.
- 65. Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, et al. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003;289(22):2983-91.
- 66. Corrigan JD. Development of a scale for assessment of agitation following traumatic brain injury. J Clin Exp Neuropsychol. 1989;11(2):261-77.
- 67. Bogner JA, Corrigan JD, Stange M, Rabold D. Reliability of the Agitated Behavior Scale. J Head Trauma Rehabil. 1999;14(1):91-6.
- 68. Buttes P, Keal G, Cronin SN, Stocks L, Stout C. Validation of the critical-care pain observation tool in adult critically ill patients. Dimens Crit Care Nurs. 2014;33(2):78-81.
- 69. Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, et al. Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011;41(6):1073-93.
- 70. McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012;22(3):276-82.
- 71. Puntillo K, Gelinas C, Chanques G. Next steps in ICU pain research. Intensive Care Med. 2017;43(9):1386-8.


# 10. Time frame and budget

Table 1. Time frame

| Month | Activities |
|---|---|
| October 2017 | - First draft of protocol |
| November 3, 2017 | - Protocol presentation to the Faculty |
| November 2017 | <ul><li>Creation of data collection sheets</li><li>Final version of research protocol</li></ul> |
| December 1, 2017 | - Research protocol submission to the Faculty |
| January 2018 | <ul> <li>Research protocol submission to the MUHC Research Ethics</li> <li>Board</li> <li>Pre-evaluation of the data collection sheets</li> <li>SPSS database creation</li> </ul> |
| January 23, 2018 | - MUHC Research Ethics Board approval |
| February to October<br>2018 | <ul> <li>Data collection</li> <li>Data entry</li> <li>Statistical analysis</li> <li>First draft of manuscript</li> </ul> |
| October 2018 | - Manuscript review |
| November 2018 | - Manuscript submission |
| December 7, 2018 | <ul> <li>Poster presentation at the Faculty (Rendez-vous de la<br/>recherche pharmaceutique)</li> </ul> |

Table 2. Budget

| Description | Туре | Total cost |
|--------------------------|-----------------|--------------------|
| Biomarker measure | Material | \$900.00 |
| Statistician (\$75.00/h) | Human resources | \$0.00 to \$200.00 |
| SPSS software | Equipment | \$0.00 |
| Paper/Poster | Material | \$200.00 |
| Total | | \$1,300.00 |

# 11. Appendices

# Appendix I. Research strategy in Medline

| Search | Terms |
|---|---|
| A1: Opioids | exp Narcotics/ or Narcotics, Pharmacological Action/ or exp Opiate Alkaloids/ or exp Fentanyl/ or exp Meperidine/ or exp Morphine Derivatives/ or exp Methadone/ or narcoti*.mp. or opioid.mp. or opium.mp. or opiate.mp. or remifentanil.mp. or fentanyl.mp. or sufentanil.mp. or alfentanil.mp. or codeine.mp. or morphine.mp. or oxycodone.mp. or hydrocodone.mp. or hydromorphone.mp. or methadone.mp. or meperidine.mp. |
| A2: Sedatives or analgesics | "Hypnotics and Sedatives"/ OR "Hypnotics and Sedatives, Pharmacological Action"/ OR Narcotics, Pharmacological Action/ OR Conscious Sedation/ OR Deep Sedation/ OR exp Narcotics/ OR exp Opiate Alkaloids/ OR exp Fentanyl/ OR exp Meperidine/ OR exp Benzodiazepines/ OR exp Morphine Derivatives/ OR exp Methadone/ OR Clonazepam/ OR Bromazepam/ OR hypnotic.mp. OR sedative.mp. OR sedation.mp. OR narcoti*.mp. OR opioid.mp. OR opium.mp. OR opiate.mp. OR remifentanil.mp. OR fentanyl.mp. OR sufentanil.mp. OR alfentanil.mp. OR codeine.mp. OR morphine.mp. OR oxycodone.mp. OR hydrocodone.mp. OR hydromorphone.mp. OR methadone.mp. OR meperidine.mp. OR benzodiazepine.mp. OR diazepam.mp. OR lorazepam.mp. OR midazolam.mp. OR clonazepam.mp. OR alprazolam.mp. OR oxazepam.mp. OR temazepam.mp. OR bromazepam.mp. OR flurazepam.mp. OR chlordiazepoxide.mp. OR clobazam.mp. OR clorazepate.mp. OR nitrazepam.mp. OR triazolam.mp. |
| B: latrogenic<br>withdrawal | Substance Withdrawal Syndrome/ OR latrogenic Disease/ OR Withholding treatment/ OR substance withdrawal.mp. OR drug withdrawal.mp. OR taper.mp. OR tapered.mp. OR tapering.mp. OR wean.mp. OR weaned.mp. OR weaning.mp. OR abstinence.mp. OR iatrogenic disease.mp. OR "withholding treatment".mp. OR "withholding treatment".mp. |
| C: ICU | exp Critical Care/ OR Subacute Care/ OR Postoperative Care/ OR exp Intensive Care Units/ OR Critical Illness/ OR intensive care.mp. OR critical care.mp. OR ICU.mp. OR PICU.mp. OR subacute.mp. OR postoperative.mp. OR postoperative.mp. OR burn unit.mp. OR burn centre.mp. OR burn center.mp. OR coronary care.mp. OR respiratory care.mp. OR critical illness.mp. OR critically ill.mp. |
| D: Tools | Decision Trees/ OR algorithms/ OR Checklist/ OR Questionnaires/ OR scale.mp. OR scaling.mp. OR score.mp. OR scoring.mp. OR tool.mp. OR checklist.mp. OR questionnaire.mp. OR instrument.mp. OR WAT.mp. OR WAT-1.mp. OR withdrawal assessment tool.mp. OR decision tree.mp. OR algorithm.mp. OR sedation withdrawal score.mp. OR "opioid and benzodiazepine withdrawal score".mp. OR OBWS.mp. OR Sophia Observation Withdrawal.mp. |
| E1: Signs and symptoms | exp "Signs and Symptoms"/ OR exp Neurological Examination/ OR Symptom Assessment/ OR exp Vital Signs/ OR Facial Expression/ OR (symptom* OR anamne* OR dysphor* OR nause* OR vomit* OR muscle ach* OR lacrim* OR rhinorrhea OR pupil* dilat* OR piloerection OR sweat* OR diarrhea OR yawn* OR fever OR temperature OR insomnia OR shiver* OR sleep disturbance OR tremor OR anxiety OR agitat* OR suction* OR irritab* OR grimac* OR startl* OR muscle tone OR |

| | ((uncoordinat* OR repetitive) AND movement) OR sneez* OR tachypnea OR |
|---|---|
| | mydriasis OR deliri* OR seiz* OR convuls*).mp. |
| E2: | exp Biomarkers/ OR "Biomarkers, Pharmacological"/ OR Monitoring, Physiologic/ OR |
| Biomarkers | Drug Monitoring/ OR Neuromuscular Monitoring/ OR Neurophysiological Monitoring/ |
| | OR (stress hormone OR cortisol OR cortisone OR catecholamines OR ((bio OR |
| | biological OR lab OR laboratory OR serum OR plasma OR endpoint? OR end- |
| | point?) ADJ (marker? OR surrogate?))).mp. |
| Run #1 (F) | A1 AND B AND C AND D AND E1 |
| Run #2 (G) | (A1 AND B AND C AND D AND E2) NOT F |
| Run #3 (H) | (A2 AND B AND C AND D AND E1) NOT (F OR G) |
| Run #4 (I) | (A2 AND B AND C AND D AND E2) NOT (F OR G OR H) |
| Run #5 (J) A1 AND B AND E2 (NOT F OR G OR H OR I) | |
| Run #6 (K) | A2 AND B AND E2 (NOT F OR G OR H OR I OR J) |

### Appendix II. Study procedure




Appendix III. Dependent variables: signs and symptoms of OIWS (4, 15, 19, 20, 24)

| Category | Signs and symptoms | Definition | Type of variable |
|---|---|---|---|
| | Agitation | During ICU hospitalization: Highest RASS score recorded in the previous 24ha according to nurse assessment b, c | Qualitative ordinal |
| | | RASS -5 to 0, 1 (restlessness) or ≥ 2 (agitation) | Qualitative ordinal |
| | | After ICU transfer to another ward: Agitated Behavior Scale (ABS) score during evaluation ≤ 21: No agitation; ≥ 22: agitation | Qualitative ordinal |
| | Anxiety | According to patient or nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| | Dysphoria | According to physician DSM-5 evaluation | Qualitative nominal (dichotomous) |
| | Fever | Highest temperature value (°C) according to nurse assessment in the previous 24h | Quantitative continuous |
| | | Temperature ≥ 38.3 degrees in the previous 24h | Qualitative nominal (dichotomous) |
| | Hallucinations | Patient seems to see, hear or feel things that are not there in the previous 24h, according to patient or nurse assessment | Qualitative nominal (dichotomous) |
| Central nervous<br>system<br>symptoms | Insomnia/sleep<br>disturbance | Number of hours of sleep/night between 10PM and 6AM the night before evaluation according to nurse assessment | Quantitative discrete |
| | | Lack of sleep defined as less<br>than 4 hours of continuous<br>sleep between 10PM and<br>6AM | Qualitative nominal (dichotomous) |
| | Startle to stimulus | Startle occurs when patient is stimulated verbally or by light touch during evaluation | Qualitative nominal (dichotomous) |
| | Time to regain calm post- | Time (minutes) needed to regain calm post-stimulus | Quantitative continuous |
| | stimulus | Normal: < 2 min; Increased: 2 to 5 min; High: > 5 min | Qualitative ordinal |
| | Seizure | Presence not explained by metabolic disturbances or history of seizures in the previous 24h according to medical chart | Qualitative nominal (dichotomous) |
| | Tremor | Presence of trembling, involuntary sustained rhythmic movements of hands and/or | Qualitative nominal (dichotomous) |

| | | feet during evaluation or | |
|---|---|---|---|
| | | according to nurse | |
| | | assessment in the previous 24h | |
| | Pupil size | Size (mm) according to nurse | Quantitative continuous |
| | . 0,0 0.20 | assessment in the previous 24h | |
| | | ≤ 2 mm, > 2 mm | Quantitative discrete |
| | | | (dichotomous) |
| | Yawning | Number of yawns in the | Quantitative continuous |
| | | previous 24h according to | |
| | | nurse assessment | O |
| | | If ≥ 2 yawns observed during | Quantitative discrete (dichotomous) |
| | | evaluation or in the previous 24h according to nurse | (dicholomous) |
| | | assessment | |
| | Hypertension | Highest Systolic blood pressure | Quantitative continuous |
| | - • | (mmHg) according to nurse | |
| | | assessment in the previous 24h | |
| | | Highest MAP (mmHg) | Quantitative continuous |
| | | according to nurse | |
| Cardiac | Tachyoardia | assessment in the previous 24h | Quantitative continuous |
| symptoms | Tachycardia | Highest HR in the previous 24h | Quantifalive Cornilloous |
| | | Lowest heart rate in previous | Quantitative continuous |
| | | 24h | |
| | | Is patient on a beta-blocker; | Qualitative nominal |
| | | Yes or No | (dichotomous) |
| | Frequent | Number of times patient | Quantitative continuous |
| | suction | required endotracheal suctioning in the previous 24h | |
| | | according to nurse | |
| | | assessment | |
| | Lacrimation | Presence during evaluation or | Qualitative nominal |
| | | according to nurse | |
| | | assessment in the previous 24h | |
| | Rhinorrhea | Presence during evaluation or | Qualitative nominal |
| | | according to nurse | (dichotomous) |
| | Sneezing | assessment in the previous 24h Number of sneeze observed | Quantitative continuous |
| Respiratory | JI IOOZII IG | during evaluation or | Qualificative continuous |
| symptoms | | according to nurse | |
| | | assessment in the previous 24h | |
| | | If more than 1 sneeze | Qualitative nominal |
| | | observed during evaluation or | (dichotomous) |
| | | according to nurse | |
| | Cianificant | assessment in the previous 24h | Ougatitative esstimates |
| | Significant dyspnea | Highest respiratory rate (RR) recorded in the previous 24h | Quantitative continuous |
| | aysprica | according to nurse | |
| | | assessment | |
| | | Lowest respiratory rate (RR) | Quantitative continuous |
| 1 | | recorded in the previous 24h | |

| | | according to nurse assessment | |
|---|---|---|---|
| | Diarrhea | Presence of ≥ 3 BMs<br>(loose/watery stools), in past<br>24 hours according to nurse<br>assessment | Qualitative nominal (dichotomous) |
| | | Number of BM in the previous 24h according to nurse assessment | Quantitative continuous |
| | | Rectal tube required (yes or no) | Qualitative nominal (dichotomous) |
| Gastrointestinal<br>symptoms | Feeding<br>intolerance<br>(gastric<br>residuals) | Present if nurse discontinued or decreased enteral feeding during previous 24h due to gastric residuals of more than 500 mL according to nurse assessment | Qualitative nominal (dichotomous) |
| | Nausea | Presence during previous 24h according to patient, nurse assessment or use of antiemetic medications such as dimenhydrinate and ondansetron (indication to validate with nurse when necessary) | Qualitative nominal (dichotomous) |
| | Vomiting | Presence or absence of vomiting episode(s) or retching or gagging in the previous 24h according to nurse assessment | Qualitative nominal (dichotomous) |
| | Mottling | Presence of violaceous marbled discoloration of the skin during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| Dermatologic<br>symptoms | Piloerection | Presence during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| | Sweating | Presence without apparent reason (not caused by room temperature) during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| | Bone, joint or<br>muscle aches | Presence during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| Musculoskeletal<br>symptoms | Muscle cramps | Presence during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |
| | Muscle tone | Presence during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |

| | (e.g. clenching wrists and toes, hunched shoulders, abnormal tense position of head, arm or legs) | |
|---|---|---|
| Uncoordinated/<br>repetitive<br>movement | Presence of involuntary movements of arm and/or legs, muscle twitches, during evaluation or according to nurse assessment in the previous 24h | Qualitative nominal (dichotomous) |

<sup>&</sup>lt;sup>a</sup> Previous 24h designate the interval between midnight of the previous day and midnight of the day on which evaluation of the signs and symptoms occurs. A fixed time frame was chosen to standardize collection of signs and symptoms.

<sup>&</sup>lt;sup>b</sup> Nurse assessment comprises written (i.e. notes in medical chart or patient flow sheet) and/or verbal communication.

<sup>&</sup>lt;sup>c</sup> On the day of transfer, patients will be evaluated from midnight of the previous day until time of evaluation. Following transfer to ward, patients will be evaluated from midnight of the current day to time of evaluation.

# Appendix IV. Diagnostic and Statistical Manual of Mental Diagnosis-V (DSM-5): "Opioid Withdrawal" criteria.

#### Diagnostic criteria:

- A. Presence of either of the following;
  - 1. Cessation of (or reduction in) opioid use that has been heavy and prolonged (i.e., several weeks or longer).
  - 2. Administration of an opioid antagonist after a period of opioid use.
- B. Three (or more) of the following developing within minutes to several days after
  - 1. Dysphoric mood.
  - 2. Nausea or vomiting.
  - 3. Muscle aches.
  - 4. Lacrimation or rhinorrhea.
  - 5. Pupillary dilation, piloerection, or sweating.
  - 6. Yawning.
  - 7. Fever.
  - 8. Insomnia.
- C. The signs or symptoms in Criterion B cause clinically significant distress or impairment in social, occupational, or other important areas of functioning.
- D. The signs or symptoms are not attributable to another medical condition and are not better explained by another mental disorder, including intoxication or withdrawal from another substance.

**Reference:** Association AP. Diagnostic and Statistical Manual of Mental Disorders: DSM-5. 5th ed. Washington, DC: American Psychiatric Publishing; 2013.


# Appendix V. Acute Physiology and Chronic Health Evaluation II (APACHE II) developed by Knaus et al.

| PHYSIOLOGIC VARIABLE | HIGH ABNORMAL RANGE | | | LOW ABNORMAL RANGE | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | +4 | +3 | +2 | +1 | 0 | +1 | +2 | +3 | +4 |
| TEMPERATURE — rectal (*C) | ≥41* | 39*-40.9* | | 38.5*38.9* | 36 - 38.4 | 34 - 35.9 - | 32.33.9. | 30*-31.9* | ≤29.9* |
| MEAN ARTERIAL PRESSURE — mm Hg | ≥ 160<br>O | 130-159 | 110-129 | | 70-109 | | 50-69 | | ≤49 |
| HEART RATE<br>(ventricular response) | O<br>≥180 | O<br>140-179 | O<br>110-139 | | O<br>70-109 | | 55-69 | O<br>40:54 | O<br>≤39 |
| RESPIRATORY RATE —<br>(non-ventilated or ventilated) | O<br>≥50 | O<br>35-49 | | O<br>25-34 | 0 | 0 | 0 | | 0 |
| OXYGENATION: A-aDO, or PaO, (mm Hg)<br>a. FiO, ≥ 0.5 record A-aDO, | O<br>≥ 500 | O<br>350-499 | O<br>200349 | | O<br><200 | | | | |
| b. FIO <sub>2</sub> < 0.5 record only PaO <sub>2</sub> | | | | | | OPO, 61-70 | | OPO, 55-60 | |
| ARTERIAL pH | ≥93 | 7.6-7.69 | | 7.5-7.59 | 7.33-7.49 | | 7.25-7.32 | 7.15-7.24 | < 7.15 |
| SERUM SODIUM (mMol/L) | ≥180 | 160-179 | 155-159 | 150-154 | 130-149 | | 120-129 | 111-119 | ≤110 |
| SERUM POTASSIUM (mMol/L) | ٥٩ | 6-6.9 | | 5.5-5.9 | 3.5-5.4 | 3-3.4 | 2.52.9 | | <2.5 |
| SERUM CREATININE (mg/100 mt)<br>(Double point score for acute renal failure) | O<br>≥3.5 | 23.4 | O<br>1.5-1.9 | | O<br>0.6-1.4 | | < 0.6 | | |
| HEMATOCRIT (%) | >0 | | 50-59.9 | 46-49.9 | 30-45.9 | | 20-29.9 | | O<br><20 |
| WHITE BLOOD COUNT (total/mm3) | 0 ≥40 | | 20-39.9 | 15-19.9 | 3-14.9 | | 1-2.9 | | ૂ |
| GLASGOW COMA SCORE (GCS):<br>Score = 15 minus actual GCS | | | | | | | | | |
| Total ACUTE PHYSIOLOGY SCORE (APS):<br>Sum of the 12 individual variable points | | | | | | | | | |
| Serum HCO, (venous-mMoVL)<br>[Not preferred, use if no ABGs] | ≥ 52 | O<br>41-51.9 | | 32.40.9 | 22-31.9 | | 18-21.9 | O<br>15-17.9 | 0 < 15 |
| as follows: sufficiency or : as follows: sufficiency or : as follows: 48.54 2 or 95.54 3 b. for elective 65.74 5 DEFINITIONS Organ Insufficients and confollows: 5.75 b. CVER: Biopsy phyperfension; c fributed to port | as a history of as immuno-comprative or emergen 5 points postoperative parency or immuno-nevident prior to the following foven cirrhosts of past a pisodes of past | and documented<br>upper GI bleeding<br>or prior episodes | oints Class RESPI vascul tion, i. duties secon sion (: te RENAI mis- IMMUI therap portal term of at that is | IOVASCULAR: N IV. RATORY: Chror ar disease resul e, unable to clir or documented dary polycythem >40mmHgl, or re: Receiving chr NO-COMPROPRESSion, recent high do sufficiently adv | nic restrictive, of<br>ting in severe en<br>bistairs or per<br>chronic hypoxi-<br>ia, severe pulmi<br>espirator depen-<br>conic dialysis.<br>ED: The patien<br>es resistance to<br>chemotherapy, it<br>se steroids, or<br>anced to suppri | bistructive, or<br>exercise restric-<br>form household<br>a, hypercapnia,<br>onary hyperten-<br>dency.<br>It has received<br>infection, e.g.,<br>adiation, long<br>as a disease<br>ass resistance to | Sum of A PS p B Age po C Chron | oints | + C : |

**Reference:** Knaus W, Draper E, Wagner D, Zimmerman J. APACHE II: a severity of disease classification system. Crit Care Med. 1985;13(10):818-29.


# Appendix VI. Glasgow Coma Scale (GCS) developed by Jennett et al.

| test | score | condition |
|---|---|---|
| | 4 | the patient can open his eyes spontaneously |
| Euo Oponina | 3 | the patient can open his eyes on verbal command |
| Eye Opening | 2 | the patient opens his eyes only in response to painful stimuli |
| 3 | 1 | the patient does not open his eyes in response to any stimulus |
| | 5 | the patient is oriented and can speak coherently |
| | 4 | the patient is disoriented but can speak coherently |
| Best Verbal<br>Response | 3 | the patient uses inappropriate words or incoherent language |
| | 2 | the patient makes incomprehensible sounds |
| | 1 | the patient gives no verbal response at all |
| | 6 | the patient can move his arms and legs in response to verbal commands |
| Best Motor<br>Response | 2-5 | the patient shows movement in response to a variety of stimuli, including pain |
| | 1 | the patient shows no movement in response to stimuli |

The results of the three tests are added up to determine the patient's overall condition

| Total score | scale |
|-------------|----------------------|
| 13-15 | mild head injury |
| 9-12 | moderate head injury |
| 3-8 | severe head injury |

Source: U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Neurological Disorders and Stroke. www.ninds.nih.gov

**Reference:** Jennett B. The Glasgow Coma Scale: History and current practice. Trauma. 2002;4(2):91-103

Appendix VII. Child-Turcotte-Pugh score developed by Pugh et al.

Table I.—GRADING OF SEVERITY OF LIVER DISEASE

| CLINICAL AND BIOCHEMICAL | POINTS SCORED FOR INCREASING<br>ABNORMALITY | | |
|---|---|---|---|
| Measurements | 1 | 2 | 3 |
| Encephalopathy (grade)* Ascites Bilirubin (mg. per 100 ml.) Albumin (g. per 100 ml.) Prothrombin time (sec. prolonged) For primary biliary cirrhosis: Bilirubin (mg. per 100 ml.) | None<br>Absent<br>1-2<br>3.5<br>1-4 | 1 and 2<br>Slight<br>2-3<br>2.8-3.5<br>4-6<br>4-10 | 3 and 4<br>Moderate<br>>3<br><2.8<br>>6<br>>10 |

<sup>\*</sup> According to grading of Trey, Burns, and Saunders (1966).

**Reference:** Pugh R, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. British Journal of Surgery. 1973 Aug 1;60(8):646-9.


# Appendix VIII. Confusion Assessment Method in the Intensive Care Unit (CAM-ICU) developed by Ely et al.

| | | Features and Descriptions | Absent | Present |
|---|---|---|---|---|
| Ī. | Acute ons | et or fluctuating course* | | |
| | <ul><li>B. Or, did<br/>and go</li></ul> | evidence of an acute change in mental status from the baseline? the (abnormal) behavior fluctuate during the past 24 hours, that is or increase and decrease in severity as evidenced by fluctuations in Sedation Scale (RASS) or the Glasgow Coma Scale? | s, tend to d | |
| II. | Inattentio | n† | | |
| | than 8 cor | tient have difficulty focusing attention as evidenced by a score of<br>rect answers on either the visual or auditory components of the A<br>Examination (ASE)? | | |
| III. | Disorgani | zed thinking | | |
| | to 3 or mo<br>Questions<br>1. Will<br>2. Are<br>3. Doo<br>4. Car<br>Commanc<br>1. Are<br>2. Hol<br>3. No<br>of t<br>(If the Ithinkin<br>unclear | a stone float on water? there fish in the sea? as 1 pound weigh more than 2 pounds? n you use a hammer to pound a nail? Is you having unclear thinking? d up this many fingers. (Examiner holds 2 fingers in front of the p. w do the same thing with the other hand (without holding the 2 fir he patient). Datient is already extubated from the ventilator, determine whethe g is disorganized or incoherent, such as rambling or irrelevant cor or or illogical flow of ideas, or unpredictable switching from subject | atient.)<br>ngers in fro<br>er the patie<br>nversation | nnt<br>nnt's |
| IV. | Altered le | vel of consciousness | | |
| | lethargic o<br>Alert:<br>Vigilant: | ent's level of consciousness anything other than alert, such as be r in a stupor, or coma? spontaneously fully aware of environment and interacts appropri hyperalert drowsy but easily aroused, unaware of some elements in the enspontaneously interacting with the interviewer; becomes fully awappropriately interactive when prodded minimally difficult to arouse, unaware of some or all elements in the enviror spontaneously interacting with the interviewer; becomes incomp prodded strongly; can be aroused only by vigorous and repeated as soon as the stimulus ceases, stuporous subject lapses back state unarousable, unaware of all elements in the environment with no interaction or avaragence of the interviewer so that the interviewer. | ately vironment are and nment or n eletely awai d stimuli ar into unresp | or not<br>ot<br>re when<br>nd<br>ponsive |
| | | interaction or awareness of the interviewer so that the interview i<br>with maximal prodding | s impossib | ile even |
| | | ICU Assessment (Features 1 and 2 and either Feature 3 or 4) | | |

unresponsive). Under the RASS system, patients who were spontaneously alert, calm, and not agitated were scored at 0 (neutral zone). Anxious or agitated patients who were sport anestus; alon, carry, are not agitated were score at 0 (neutral zone). Anxious or agitated patients received a range of scores depending on their level of anxiety: 1 for anxious, 2 for agitated (fighting ventilator), 3 for very agitated (pulling on or removing catheters), or 4 for combative (violent and a danger to staff). The scores –1 to –5 were assigned for patients with varying degrees of sedation based on their ability to maintain eye contact: –1 for more than 10 seconds, –2 for less than 10 seconds, and –3 for eye opening but no eye contact. If physical stimulation was required, then the patients were scored as either –4 for eye opening or movement with physical or painful stimulation or -5 for no response to physical or painful stimulation. The RASS has excellent interrater reliability and intraclass correlation coefficients of 0.95 and 0.97, respectively, and has been validated against visual analog scale and geropsychiatric diagnoses in 2 ICU studies. 97.50 †In completing the visual ASE, the patients were shown 5 simple pictures (previously published<sup>54</sup>) at 3-second intervals

letters from the following list in a normal tone at a rate of 1 letter per second: S, A, H, E, V, A, A, R, A, T. A scoring method similar to that of the visual ASE was used for the auditory ASE testing.

This table may be reproduced without permission for clinical use only (Ely EW et al. JAMA. 2001;286:2707-2710).

Reference: Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, et al. Delirium in mechanically ventilated patients; validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). Jama. 2001;286(21):2703-10.

# Appendix IX. Confusion Assessment Method (CAM) developed by Inouye et al.

# Appendix Table 1. The Confusion Assessment Method Instrument Acute onset 1. Is there evidence of an acute change in mental status from the patient's baseline? A. Did the patient have difficulty focusing attention, for example, being easily distractible, or having difficulty keeping track of what was being said? Not present at any time during interview. Present at some time during interview, but in mild form. Present at some time during interview, in marked form. Uncertain. B. (If present or abnormal) Did this behavior fluctuate during the interview, that is, tend to come and go or increase and decrease in severity? No. Uncertain Not applicable. C. (If present or abnormal) Please describe this behavior: 3. Was the patient's thinking disorganized or incoherent, such as rambling or irrelevant conversation, unclear or illogical flow of ideas, or unpredictable switching from subject to subject? Altered level of consciousness 4. Overall, how would you rate this patient's level of consciousness? Alert (normal). Vigilan (hyperalert, overly sensitive to environmental stimuli, startled very easily). Letharpic (drowsy, easily aroused). Supor (difficult to arouse). Coma (unarousable). Uncertain. 5. Was the patient disoriented at any time during the interview, such as thinking that he or she was somewhere other than the hospital, using the wrong bed, or misjudging the time of day? 6. Did the patient demonstrate any memory problems during the interview, such as inability to remember events in the hospital or difficulty remembering instructions? Perceptual disturbances Did the patient have any evidence of perceptual disturbances, for example, hallucinations, illusions, or misinterpretations (such as thinking something was moving when it was not)? At any time during the interview, did the patient have an unusually increased level of motor activity, such as restlessness, picking at bedelothes, tapping fingers, or making frequent sudden changes of position? At any time during the interview, did the patient have an unusually decreased level of motor activity, such as sluggishness, staring into space, staying in one position for a long time, or moving very slowly?

#### Appendix Table 2. The Confusion Assessment Method (CAM) Diagnostic Algorithm\*

\* The questions listed under this topic were repeated for each topic where applicable

#### Feature 1. Acute Onset and Fluctuating Course

This feature is usually obtained from a family member or nurse and is shown by positive responses to the following questions: Is there evidence of an acute change in mental status from the patient's baseline? Did the (abnormal) behavior fluctuate during the day, that is, tend to come and go, or increase and decrease in severity?

 Did the patient have evidence of disturbance of the sleep-wake cycle, such as excessive daytime sleepiness with insomnia at night?

#### Feature 2. Inattention

This feature is shown by a positive response to the following question: Did the patient have difficulty focusing attention, for example, being easily distractible, or having difficulty keeping track of what was being said?

#### Feature 3. Disorganized Thinking

This feature is shown by a positive response to the following question: Was the patient's thinking disorganized or incoherent, such as rambling or irrelevant conversation, unclear or illogical flow of ideas, or unpredictable switching from subject to subject?

#### Feature 4. Altered Level of Consciousness

This feature is shown by any answer other than "alert" to the following question: Overall, how would you rate this patient's level of consciousness? (alert [normal], vigilant [hyperalert], lethargic [drowsy, easily aroused], stupor [difficult to arouse], or coma [unarousable])

**Reference:** Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: The confusion assessment methoda new method for detection of delirium. Annals of internal medicine. 1990 Dec 15;113(12):941-8


<sup>\*</sup> The diagnosis of delirium by CAM requires the presence of features 1 and 2 and either 3 or 4.

## Appendix X. Richmond Agitation-Sedation Scale (RASS) developed by Sessler et al.

| Score | Term | Description |
|---|---|---|
| +4 | Combative | Overtly combative or violent; immediate danger to staff |
| +3 | Very agitation | Pulls on or removes tube(s) or catheter(s) or has aggressive behavior<br>toward staff |
| +2 | Agitated | Frequent nonpurposeful movement or patient-ventilator dyssynchrony |
| +1 | Restless | Anxious or apprehensive but movements not aggressive or vigorous |
| 0 | Alert and calm | |
| -1 | Drowsy | Not fully alert, but has sustained (more than 10 seconds) awakening, with eye contact, to voice |
| -2 | Light sedation | Briefly (less than 10 seconds) awakens with eye contact to voice |
| -3 | Moderate sedation | Any movement (but no eye contact) to voice |
| -4 | Deep sedation | No response to voice, but any movement to physical stimulation |
| -5 | Unarousable | No response to voice or physical stimulation |

#### Procedure

- Observe patient. Is patient alert and calm (score 0)?
   Does patient have behavior that is consistent with restlessness or agitation (score +1 to +4 using the criteria listed above, under excessive).
- If patient is not alert, in a loud speaking voice state patient's name and direct patient to open eyes and look at speaker. Repeat once if necessary. Can prompt patient to continue looking at speaker.
  - Patient has eye opening and eye contact, which is sustained for more than 10 seconds (score -1).
  - Patient has eye opening and eye contact, but this is not sustained for 10 seconds (score -2).
  - Patient has any movement in response to voice, excluding eye contact (score -3).
- If patient does not respond to voice, physically stimulate patient by shaking shoulder and then rubbing sternum if there is no response to shaking shoulder.
  - Patient has any movement to physical stimulation (score -4).
  - Patient has no response to voice or physical stimulation (score -5).

**Reference:** Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, et al. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002;166(10):1338-44.

# Appendix XI. Agitated Behavior Scale (ABS) developed by Carrigan et al.

# AGITATED BEHAVIOR SCALE

| Patient | | Period of | Observatio | nn. | |
|---|---|---|---|---|---|
| - uncin | | I cilou oi | a.m. | <b>J11.</b> | |
| Observ | Environ | From | p.m | 1 | 1 |
| ODSCIV. | Litviron. | 110111 | p.m<br>a.m. | | |
| Rater/Di | sc. | To: | | / | |
| each iten | nd of the observation period in was present and, if so, to woollowing numerical values a | hat degree: sligh | it, moderat | | |
| $2 = p_1$ $3 = p_1$ $4 = p_1$ | psent: the behavior is not pro-<br>resent to a slight degree: the<br>the conduct of other, contexts<br>may redirect spontaneously,<br>does not disrupt appropriate<br>resent to a moderate degree:<br>an agitated to an appropriate<br>resent to an extreme degree:<br>appropriate behavior due to<br>even when external cueing of | e behavior is presually appropriate or the continuation behavior. ) the individual nebehavior, but be the individual is the interference of | e behavior.<br>on of the ag<br>needs to be<br>enefits from<br>a not able to<br>of the agitat | (The gitated redire such o enga | individual<br>d behavior<br>cted from<br>cueing.<br>ige in |
| DONO | T LEAVE BLANKS. | | | | |
| 1. | Short attention span, easy o | listractibility, ina | bility to co | ncentr | ate. |
| 2. | Impulsive, impatient, low t | olerance for pain | or frustrat | ion. | |
| 3. | Impulsive, impatient, low t<br>Uncooperative, resistant to<br>Violent and or threatening | care, demanding | <b>5.</b> | | |
| 4. | Violent and or threatening | violence toward | people or p | roper | t <del>y</del> . |
| 5. | Explosive and / or unpredic | table anger. | | | |
| 6. | Rocking, rubbing, moaning | or other self-stin | nulating be | havio | r. |
| 7. | Pulling at tubes, restraints,<br>Wandering from treatment<br>Restlessness, pacing, excess | etc. | | | |
| 8. | Wandering from treatment | areas. | | | |
| 9. | Restlessness, pacing, excess | ive movement. | | | |
| 10. | Repetitive behaviors, motor | r and/or verbal. | | | |
| 11. | Rapid, loud or excessive tal | king. | | | |
| 12. | Sudden changes of mood. | | 1. | | |
| 13. | Easily initiated or excessive | crying and/or la | aughter. | | |
| 14. | Self-abusiveness, physical a | ind/or verbal. | | | |

**Reference:** Corrigan JD. Development of a scale for assessment of agitation following traumatic brain injury. Journal of Clinical and Experimental Neuropsychology. 1989 Mar 1;11(2):261-77.


\_\_\_\_ Total Score

Appendix XII. Critical-Care Pain Observation Tool (CPOT) developed by Gelinas et al.

| Indicator | Score | | Checklist |
|---|---|---|---|
| Facial expression | Relaxed, neutral | 0 | No muscle tension observable Eyes closed |
| | Tense | 1 | Frowning/Brow lowering Orbit tightening/Wincing Levator contraction Mouth opening Eye opening Eye weeping/tears Eyebrow raising Blinking |
| | Grimacing | 2 | Frowning/Brow lowering Eyes tightly closed Levator contraction Mouth opening Biting endotracheal tube/Clenched teeth Flushing |
| Body movements | Absence of movements or normal position | 0 | Does not move at all □<br>Normal position □ |
| | Protection | 1 | Slow, cautious movements Limb flexion Trying to reach pain site/tubes Touching pain site/Guarding Seeking attention Rubbing/Massaging pain site Shaking Withdrawing Decortication Decerebration |
| | Restlessness/Agitation | 2 | Touching/Pulling tubes Fidgeting/Restlessness Arching Pushing Striking at staff/Defensive grabbing Attempting to sit up Trying to climb out of bed |
| Compliance with the ventilator (intubated patients) | Tolerating ventilator or movement Coughing but tolerating | 0 | Alarms not activated, easy ventilation Alarms activated, stop spontaneously Coughing Gag reflex |
| OR | Fighting ventilator | 2 | Asynchrony □ Blocking ventilation □ |
| Vocalization (extubated patients) | Talking in normal tone or no sound | 0 | No sound □ Normal tone □ |
| | Sighing, moaning | 1 | Sighing □ Moaning □ Verbal complaints of pain □ |
| | Crying out, sobbing | 2 | Crying out □ Sobbing □ |
| Muscle tension | Relaxed | 0 | No resistance to passive movements |
| Evaluation by passive flexion and extension of upper limbs when | , , | 1 | Resistance to passive movements |
| patient is at rest or evaluation when patient is being turned | Very tense or rigid | 2 | Strong resistance to passive movements Clenching fists |
| TOTAL | /8 | | |

**Reference:** Gelinas C, Fillion L, Puntillo K, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006;15(4):420-7.


# Appendix XIII. Numeric Rating Scale (NRS)

| Numerical rating scale | |
|-------------------------------|----|
| No pain Worst imaginable pain | |
| 0 1 2 3 4 5 6 7 8 9 10 | 10 |

**Reference:** Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. Journal of clinical nursing. 2005 Aug 1;14(7):798-804.
